CLINICAL TRIAL: NCT06957860
Title: Septal Bone Expansion Using Osseodensification Versus Piezoelectric Implant Site Preparation for Immediate Implant Placement in Mandibular Molars [Randomized Clinical Trial]
Brief Title: Septal Bone Expansion Using Osseodensification Versus Piezoelectric Implant Site Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0716-06/2023
Record Dates: First submitted 2025-04-27; First posted 2025-05-05 (Actual); Last update posted 2025-05-05 (Actual); Status verified 2025-04

CONDITIONS: Dental Implant; Osseodensification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the statistician will be blinded to the treatment groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- piezoelectric group (Experimental)
  Interventions: Other: Piezotome
- osseodensification (Experimental)
  Interventions: Other: Densah burs

INTERVENTIONS:
Other: Piezotome — Four Intra-lift diamond tips were used for drilling the osteotomy, increasing diameters till a final diameter of 2.8 mm is reached for placement of 3.5 mm diameter and 10-12 mm length implant.
  Arms: piezoelectric group
Other: Densah burs — implant drilling procedures will be done using the surgical drills of the supplier kit of densah burs. Surgical drills of increasing diameters will be used till a final drill diameter of 3 mm for placement of a 3.5 mm diameter.
  Arms: osseodensification

SUMMARY:
: Implant placement in the inter radicular septum is usually considered the best option for an immediate molar implant, not only in terms of correct 3D positioning, but also regarding implant survival, Osseodensification was shown to enhance implant primary stability, due to the compaction auto-grafting and the associated spring-back effect. Piezoelectric implant site preparation (PISP) has been proposed as an alternative technique to improve surgical control, safety, and bone healing response Aim of the work: To evaluate and compare stability changes using insertion torque values (ITV) and Implant Stability Quotient values (ISQ) for immediately placed implants in molar septum using Osseodensification technique and Piezoelectric implant site preparation (PISP) technique.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hopeless mandibular molar teeth in the posterior region in need of implant placement .
* A fully intact facial bone wall at the extraction site.
* Systemically healthy, received no head and neck radiation for cancer treatment.
* Absence of periapical pathologies or suppuration at the time of installing the implants.
* Septal bone after atraumatic extraction not less than 3 mm.

Exclusion Criteria:

* Systemic conditions that would prevent successful healing or implant osseointegration; examples are uncontrolled Diabetes Mellitus, metabolic bone disorders, autoimmune diseases, or Bisphosphonate therapy.
* Heavy smoker patients.
* Presence of preapical bone loss related to extracted tooth.
* Patient is not indicated for immediate implant placement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Change in implant stability | Baseline and 3 months
  The implant stability quotient (ISQ) will be measured using the Osstell device- resonance frequency analysis test at 3 months post-surgery to all the installed fixtures.

SECONDARY OUTCOMES:
Change in bone density | Baseline and 3 months
  Using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt